CLINICAL TRIAL: NCT04778163
Title: The Use of Humor With Young Adults in Psychiatric Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Cédric DEVILLE, Medical Doctor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDEVILLE
Record Dates: First submitted 2021-01-30; First posted 2021-03-02 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Treatment Adherence and Compliance; Psychiatric Disorder
Keywords: Young people; Young adults; Humor; Psychotherapy; Group psychotherapy; Resilience
MeSH Terms: conditions — Treatment Adherence and Compliance; Mental Disorders | interventions — Therapeutics; Psychotherapy, Group

STUDY DESIGN:
Intervention Model Description: A treatment arm receives a psychotherapeutic group intervention (based on humor with cognitive behavioural and psychoeducative approaches) over a period 6 weeks.
  A control arm is placed on a 6 week waiting list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Humor group 1 (Experimental): Group 1 - experimental - will participate in a "humor group" with a one-hour group session per week for 6 weeks.
  Interventions: Behavioral: Clinical use of humor
- Control group 2 (No Intervention): Group 2 - the control group - will follow an usual treatment regimen for 6 weeks. At the end of the "Humor Group" of group 1, the 2 groups of patients will undergo a second series of tests identical to those of the pregroup. The paired patients should be randomly assigned. The control group will do the "Humor Group" after 6 weeks.

INTERVENTIONS:
Behavioral: Clinical use of humor — Clinical study in psychiatry in young adult patients between 18 and 25 years old. The aim of the study is to evaluate the therapeutic impact of the clinical use of humor through 6 group sessions (group of 5 to 10 patients), at the rate of one hour session per week for 6 weeks.
  The investigators will form 2 groups of 5 to 10 patients matched in terms of gender, education level and score on a scale measuring their sense of humor. The participants will be asked to complete a series of tests measuring their ability to use humor, psychiatric symptoms and well-being.
  Other Names: Treatment; Group psychotherapy
  Arms: Humor group 1

SUMMARY:
Clinical study in psychiatry in young adult patients between 18 and 25 years old. The aim of the study is to evaluate the therapeutic impact of the clinical use of humor through 6 group sessions (group of 5 to 10 patients), at the rate of one hour session per week for 6 weeks.

The investigators will form 2 groups of 5 to 10 patients matched in terms of gender, education level and score on a scale measuring their sense of humor. The participants will be asked to complete a series of tests measuring their ability to use humor, psychiatric symptoms and well-being.

Group 1 (test group) will participate in the humor-based sessions, while Group 2 (control group) will receive regular treatment for 6 weeks (waiting list: patients in Group 2 will attend humor-based sessions once Group 1 has completed their 6 weeks).

At the end of the 6-week sessions, both groups will receive the same series of pre-session tests to see whether or not there has been improvement in their overall functioning, psychiatric symptomatology and appreciation/use of humor.

At the end of the 2x 6-week sessions, group 2 will again receive this series of pre-session tests to see whether or not their overall functioning, psychiatric symptomatology and appreciation/use of humour has improved.

Objective(s)/Aim:

To evaluate the resilience of young adult psychiatric patients and their ability to cope with stress through the use of humor in a set of 6 modules on the use of humor.

To evaluate the symptoms.

Outcome/Endpoints :

Using scales, measure this evolution.

DETAILED DESCRIPTION:
Project design and procedures :

The investigators will form 2 groups of 5 to 10 patients matched on their score on the sense of humor scale, their gender and their level of education. The participants will be asked to complete a series of tests measuring their ability to use humor, clinical variables and general functioning.

Group 1 - experimental - will participate in a "humor group" with a one-hour group session per week for 6 weeks.

Group 2 - the control group - will follow a usual treatment regimen for 6 weeks. At the end of the "Humor Group" of group 1, the 2 groups of patients will undergo a second series of tests identical to those of the pregroup. The paired patients should be randomly assigned. The control group will do the "Humor Group" after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Young adult patients of a psychiatric's unit (young people from 18 to 25 years old with beginner psychic disorders) who are French-speaking and able to give their informed consent.

Exclusion Criteria:

* Those who do not meet the above criteria.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Primary outcome is sense of humor using scale : Sense of Humor Scale (from 36 to 144 : higher scores mean a better outcome). | About three years
  To evaluate whether or not their appreciation/use of humor has improved.

SECONDARY OUTCOMES:
Coping evolution using scale : Coping Humor Scale (from (-14) to (+14) : higher scores mean a better outcome). | About three years
  To evaluate whether or not the coping evolution has improved.
Psychiatric symptoms evolution using scale : Brief Psychiatric Rating Scale (from 24 to 168 : higher scores mean a worse outcome). | About three years
  To evaluate whether or not the overall psychiatric symptomatology has improved.
Global functioning using scales : Global Assessment Functioning (from 1 to 100 : higher scores mean a better outcome). | About three years
  To evaluate whether or not the overall functioning has improved.
Clinical global impression using scale : Clinical Global Impression (from 1 to 7 : higher scores mean a worse outcome). | About three years
  To evaluate whether or not the overall global clinical impression has improved.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric AM Devillé, Dr, Principal Investigator — University Hospital, Geneva
Locations (1):
- Programme JADE, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bozikas VP, Kosmidis MH, Giannakou M, Anezoulaki D, Petrikis P, Fokas K, Karavatos A. Humor appreciation deficit in schizophrenia: the relevance of basic neurocognitive functioning. J Nerv Ment Dis. 2007 Apr;195(4):325-31. doi: 10.1097/01.nmd.0000243798.10242.e2. PMID 17435483
- [Background] Compas BE, Connor-Smith JK, Saltzman H, Thomsen AH, Wadsworth ME. Coping with stress during childhood and adolescence: problems, progress, and potential in theory and research. Psychol Bull. 2001 Jan;127(1):87-127. PMID 11271757
- [Background] Corcoran R, Cahill C, Frith CD. The appreciation of visual jokes in people with schizophrenia: a study of 'mentalizing' ability. Schizophr Res. 1997 Apr 11;24(3):319-27. doi: 10.1016/s0920-9964(96)00117-x. PMID 9134592
- [Background] Corrigan PW, Powell KJ, Fokuo JK, Kosyluk KA. Does humor influence the stigma of mental illnesses? J Nerv Ment Dis. 2014 May;202(5):397-401. doi: 10.1097/NMD.0000000000000138. PMID 24727719
- [Background] Franzini LR. Humor in therapy: the case for training therapists in its uses and risks. J Gen Psychol. 2001 Apr;128(2):170-93. doi: 10.1080/00221300109598906. PMID 11506047
- [Background] Valentine L, Gabbard GO. Can the use of humor in psychotherapy be taught? Acad Psychiatry. 2014 Feb;38(1):75-81. doi: 10.1007/s40596-013-0018-2. PMID 24430586
- [Background] Ventura J, Nuechterlein KH, Subotnik KL, Gutkind D, Gilbert EA. Symptom dimensions in recent-onset schizophrenia and mania: a principal components analysis of the 24-item Brief Psychiatric Rating Scale. Psychiatry Res. 2000 Dec 27;97(2-3):129-35. doi: 10.1016/s0165-1781(00)00228-6. PMID 11166085
- [Background] Derouesne C. [Neuropsychology of humor: an introduction Part 1. Psychological data]. Geriatr Psychol Neuropsychiatr Vieil. 2016 Mar;14(1):95-103. doi: 10.1684/pnv.2016.0583. French. PMID 27005341
- [Background] Etienne E, Braha S, Januel D. [Humour and the theory of mind in schizophrenia: a review of the literature]. Encephale. 2012 Apr;38(2):164-9. doi: 10.1016/j.encep.2011.03.008. Epub 2011 Jul 5. French. PMID 22516275
- [Background] McGhee, P. (1994). How to develop your sense of humor. Dubuque: Kendall Hunt.
- [Background] Rengade, C.E. (2014). L'humour en thérapie cognitive et comportementale. J thér comport cogn, 24(1), 1-4.
- [Background] Salameh, W.A. (1983). Humor in psychotherapy: past outlooks, present status, and future frontiers. In: McGhee, P.E., Goldstein, J.H., editors. Handbook of humor research. Volume II Applied studies. New York: Springer, 61-88.
- [Background] Ventura, J., Green, M.F., Shaner, A., Liberman, R.P. (1993). Training and quality assurance with the Brief Psychiatric Rating Scale: "The drift busters". International Journal of Methods in Psychiatry Research, 3, 221-224.
- [Result] Cai C, Yu L, Rong L, Zhong H. Effectiveness of humor intervention for patients with schizophrenia: a randomized controlled trial. J Psychiatr Res. 2014 Dec;59:174-8. doi: 10.1016/j.jpsychires.2014.09.010. Epub 2014 Sep 19. PMID 25266473
- [Result] Falkenberg I, Buchkremer G, Bartels M, Wild B. Implementation of a manual-based training of humor abilities in patients with depression: a pilot study. Psychiatry Res. 2011 Apr 30;186(2-3):454-7. doi: 10.1016/j.psychres.2010.10.009. Epub 2010 Nov 11. PMID 21071099
- [Result] Rudnick A, Kohn PM, Edwards KR, Podnar D, Caird S, Martin R. Humour-related interventions for people with mental illness: a randomized controlled pilot study. Community Ment Health J. 2014 Aug;50(6):737-42. doi: 10.1007/s10597-013-9685-4. Epub 2013 Dec 12. PMID 24337476
- See also: Association for Applied and Therapeutic Humor — http://www.aath.org/